CLINICAL TRIAL: NCT04437836
Title: Evaluation of Pharmacokinetics and Safety Tolerability of Higher Doses of Rifampicin in Children With Newly Diagnosed Uncomplicated Tuberculosis
Brief Title: Evaluation of Pharmacokinetics and Safety Tolerability of Higher Doses of Rifampic
Acronym: HighRif C
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kilimanjaro Clinical Research Institute (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TMA2017CDF-1876-HighRif C
Record Dates: First submitted 2020-05-28; First posted 2020-06-18 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2023-12

CONDITIONS: Clinical Trial
Keywords: Tuberculosis, Pharmacokinetics, safety/torelability
MeSH Terms: conditions — Tuberculosis | interventions — Rifampin; Clinical Trials Data Monitoring Committees

STUDY DESIGN:
Intervention Model Description: Safety and tolerability study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Enroll children participant and giving them treatment care as well as safety monitoring
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control arm (Experimental): Participants will receive standard treatment of rifampicin
  Interventions: Drug: Evaluation of high dose rifampicin in children
- First High dose (Experimental): Participants will receive 30mg per kg body weight of rifampicin
  Interventions: Drug: Evaluation of high dose rifampicin in children
- Second high dose (Experimental): Particpants will receive 40mg per kg body weight of rifampicin
  Interventions: Drug: Evaluation of high dose rifampicin in children

INTERVENTIONS:
Drug: Evaluation of high dose rifampicin in children — Evaluation of severity of adverse event from grade 1 to 5
  Other Names: Safety monitoring

SUMMARY:
Tuberculosis in children is a major public health problem and it contributes 10% of the total TB cases worldwide. TB treatment outcomes in children are challenged by insufficient consideration of the relationships between doses administered, concentrations achieved and eventual desirable and undesirable effects (pharmacodynamics) of TB drugs. Rifampicin is a pivotal TB drug and data from adults suggest that a much higher dose of rifampicin (35 mg/kg instead of 10 mg/kg), resulting in much higher rifampicin exposures in plasma, is safe and tolerable and may provide a higher efficacy. The dose needed in children to achieve the same exposure in plasma is unknown.

DETAILED DESCRIPTION:
Tuberculosis (TB) in children is a major public health problem . It has a global estimate of >100,000 deaths per year and is included in the top ten causes of mortality in children worldwide. Children contribute 10% of the total TB cases worldwide. More than 75% of the worldwide estimated cases of TB in children occur in the 30 high burden countries, Tanzania being one of them. The enormous burden of pediatric TB in these countries is due to the TB epidemic amongst adults and the simultaneous HIV pandemic and a child less than 14 years of age whether HIV infected or not is at a high risk of developing the disease. Subsequent dissemination of the mycobacterium and progression of the disease is also fast in children.

Knowledge on the efficacy and safety of medicines for children is still very limited and sometimes children are still being treated as small adults. However, adult dosing cannot be logically extrapolated to children according to weight or age because of different pharmacokinetics, i.e. the relationship between doses administered and exposures (drug concentrations) achieved, in children as compared with adults . More specifically, these pharmacokinetic differences occur in the subsequent processes of absorption, distribution, metabolism and elimination of drugs, which are subject to physiological changes due to growth and development in children. Especially in young children, maturation of liver metabolism pathways and renal function are not completed.

In contrast, the pharmacodynamics of a drug, i.e. the relationship between concentrations achieved and eventual response is generally considered similar between adults and children, although differences in drug metabolism between children and adults may lead to differences in susceptibility to some adverse drug reactions. Thus, because of the differences in pharmacokinetics in children with different ages, they should not receive the same drug doses on mg/kg base as adults, and drug dosage selection in children should rather be based upon stages of growth and development. These drug doses should target the exposures that are efficacious in adults.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 to 14 years with newly diagnosed Tuberculosis

Exclusion Criteria:

* Children with elevated liver function
* Children allergic to first line anti-TB drugs

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of high dose rifampicin | 54 months
  To know the maximum tolerable dose of rifampicin in children aged 1-14 years

SECONDARY OUTCOMES:
Plasma concentration | 54 months
  Maximum observed concentration
Time | 54 months
  To measure time to reach maximum concentration

CONTACTS AND LOCATIONS:
Locations (4):
- Tanzania (4):
  - Kilimanjaro Clinical Research Institute, Moshi, Kilimanjaro
  - Hydom Hospital, Babati, Manyara Region
  - Mt. Meru Hospital, Arusha
  - Huruma Hospital, Moshi